CLINICAL TRIAL: NCT06812819
Title: Effect of Cryostimulation on Selected Motor Skills in Soccer Players
Status: Approved for marketing | Type: Expanded Access
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Izabela Różycka, Principal Investigator, Poznan University of Physical Education
Other Study IDs: 12622001541796, ANZCTR
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Particularly Partial-body Cryostimulation
Keywords: cryotherapy; cold exposure; motor skills; soccer players; athletic recovery

INTERVENTIONS:
Diagnostic Test: Cryostimulation is a form of cooling the body using low temperatures without causing tissue damage. The stimulus effect is achieved at temperatures below - 110⁰C, in a short time of 1-3 minutes. The p — PBC protocol involved the participant being in a JUKA cryosauna (model 0104-1), for 3 minutes at - 140 ° C± - 20 ° C with the lid at shoulder height and the head over the chamber. The cryosauna was cooled with liquid nitrogen, and the temperature was monitored by a computer. Participants entered the cabin wearing clogs, wool socks, shorts, gloves, caps, and disposable PP non-woven masks to protect against inhalation of nitrogen fumes. The temperature inside the cryosauna was recorded at 30-second intervals using a sensor placed on the bottom of the cabin. The temperature of the room where the cryosauna was located was 21.0 ± 0.9° C, and the humidity of the air during the treatment was 35 ± 2, 0 % monitored with a QUIGG type LE 2014.14 moisture absorber.
  Other Names: OptoGait optical system (MicroGate Timing and Sport, BONZAMO, Italy; Tanita BC-418 MA analyzer, (Medizin & Service GmbH, Germany; JUKA cryosauna 0104-1, Germany

SUMMARY:
A randomized study was conducted during two training periods. The first stage of a 5-day cryostimulation procedure took place in November 2022, during the training period after the end of the league season. The second stage was conducted in January 2023, during the preparation period in full training loads. The sequence of procedures used in both stages was the same (fig. 1). Before the application of cryostimulation, both PBC and CON groups underwent measurements: anthropometric using Tanita BC-418 MA analyzer (Medizin & Service GmbH, Germany), step frequency (tapping) and lower limb maximal power (jump with sweep, jump without sweep), Opto Gait optical system (MicroGate Timing and Sport, BONZAMO, Italy ). Athletes in the PBC group, at the same hours of 8: 00 (stage I) and 17:00 (stage II), were subjected daily to cryostimulation in a JUKA cryosauna (model 0104-1, Germany). Both PBC and CON groups participated in training together throughout the study period.

DETAILED DESCRIPTION:
Anthropometric measurements Using Tanita BC-418 MA analyzer, (Medizin & Service GmbH, Germany), measurement accuracy was ± 0.1 kg. The following parameters were analyzed: body mass index (BMI), total body water (TBW), fat mass (FM), and fat-free mass (FFM), and basal metabolism (BMR), Table 1. All measurements were taken fasting at 8:00 a.m. on the first and fifth day of the study in both groups of subjects. The device was calibrated before each testing session according to the manufacturer's guidelines.

Fitness tests Measurements of step frequency and maximal power [W/kg] of the lower limbs were performed using the OptoGait optical system (MicroGate Timing and Sport, BONZAMO, Italy). The measurement system consisted of two panels used to detect spatial parameters for gait, jumping, and reaction time. Measurement strips were placed in parallel on the ground at a distance of 1.5 meters from each other. The test consisted of 3 parts: tapping (step frequency), maximal jumping up without upper limb sweep, and maximal jump up with upper limb assisted sweep (analysis of lower limb maximal power and jump height). Test subjects were positioned between the slats in the starting position, and performed 3 test trials, each trial began and ended with an audible signal, and the time of a single trial was 10 seconds. Analysis of the components of lower limb maximal power and step frequency was performed in the PBC and CON groups on the first and last days of the study.

Cryostimulation (PBC) PBC protocol involved the participant being in a JUKA cryosauna (model 0104-1), for 3 minutes at - 140 ° C± - 20 ° C with the lid at shoulder height and the head over the chamber. The cryosauna was cooled with liquid nitrogen, and the temperature was monitored by a computer. Participants entered the cabin wearing clogs, wool socks, shorts, gloves, caps, and disposable PP non-woven masks to protect against inhalation of nitrogen fumes. The temperature inside the cryosauna was recorded at 30-second intervals using a sensor placed on the bottom of the cabin. The temperature of the room where the cryosauna was located was 21.0 ± 0.9° C, and the humidity of the air during the treatment was 35 ± 2, 0 % monitored with a QUIGG type LE 2014.14 moisture absorber. All participants received instructions on proper breathing and cryosauna behavior before the PBC procedure. They received information on risks, complications, and indications for immediate discontinuation of the therapy. Athletes signed an informed consent for the experiment. During the PBC, they remained in constant visual and auditory contact with the therapy supervisor. A cryostimulation session was performed every day from 8:00-9:00 am, for 5 days. During one PBC treatment, the athletes spent 3 minutes at -140° C ± 20° C. Each entry into the cryosauna was preceded by a measurement of saturation temperature and blood pressure. These measurements were taken again each day immediately after exiting the cryosauna. After completing the cryotherapy procedure, the athletes were subjected to a 15-minute warm-up according to a set schedule.

ELIGIBILITY:
Inclusion Criteria:

* TraAge: 18-35 years,
* Training: at least three years,
* regular training
* Health status: no musculoskeletal injuries,
* Medical certificate from a certified sports physician indicating readiness to participate in intensive training and cryostimulation treatments.
* Lifestyle restrictions:

agreement to refrain from additional regenerative therapies, cosmetic treatments, alcohol, stimulants and dietary supplements during the study.

1. Inclusion Criteria:

   * TraAge: 18-35 years,
   * Training: at least three years, regular training
   * Health status: no musculoskeletal injuries,
   * Medical certificate from a certified sports physician indicating readiness to participate in intensive training and cryostimulation treatments.
   * Lifestyle restrictions: restrictions on additional regenerative therapies, cosmetic procedures, alcohol, stimulants and dietary supplements during the study.
2. Exclusion criteria:

   * Age: under 18 or over 35 years of age,
   * Training: less than three years of regular professional soccer training or playing.
   * Health conditions: acute or chronic injuries, cardiovascular diseases, respiratory diseases or conditions that contraindicate cryostimulation,
   * Failure to follow: planned training, testing or cryostimulation protocols; failure to follow lifestyle restrictions as outlined in the study guidelines,
   * Contraindications to cryostimulation: sensitivity or adverse reactions to cold exposure.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — technical skills (dribbling, passing, shooting), physical attributes (speed, endurance, strength), tactical awareness (positioning, game intelligence), and mental qualities (discipline, teamwork, resilience),Body structure, physical predispositions, and hormonal variability play a key role in a footballer's performance.

CONTACTS AND LOCATIONS:
Overall Officials: Izabela Różycka, mgr, Principal Investigator — Department of Physiotherapy, Poznań University of Physical Education, Faculty of Sport Sciences In Gorzów Wielkopolski; Poland
Locations (1):
- Department of Physiotherapy, Poznań University of Physical Education, Faculty of Sport Sciences In Gorzów Wielkopolski; Poland, Gorzów Wielkopolski, Lubusz Voivodeship, Poland